CLINICAL TRIAL: NCT04330417
Title: Bidirectional Myoelectric (BIMYO) Soft Robotic Glove Technology For Robot-Assisted Hand Therapy in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018/01258
Record Dates: First submitted 2019-04-24; First posted 2020-04-01 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Stroke
Keywords: Stroke; Soft Robotic Glove; Electromyography; Hand Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMG Glove Group (Experimental): A total of 12 sessions of robot-assisted hand training for 6 consecutive weeks.
  Interventions: Device: Robot-Assisted Hand Training
- Control Group (Active Comparator): A total of 12 session of standard hand therapy sessions in 6 consecutive weeks.
  Interventions: Other: Standard Hand Therapy

INTERVENTIONS:
Device: Robot-Assisted Hand Training — Perform activities of daily living, e.g., write sentences, turn cards, move small and big objects, simulated feeding, stack checkers, pour water, squeeze handles
  Arms: EMG Glove Group
Other: Standard Hand Therapy — Stretching, Strengthening, Hand Functional Training
  Arms: Control Group

SUMMARY:
Stroke patients have limited hand mobility post-stroke, thus inhibiting them from performing daily functional tasks independently, resulting in reduced quality of life. Current hand rehabilitation robotic devices are typically driven by rigid linkages/joints, which subject the fingers into a single plane of motion that is unnatural and uncomfortable. These devices belong to the class of continuous passive motion (CPM) devices that only promote hand range-of-motion, but do not require the patient to play an active role in performing the hand exercises. There is a strong need for a device that can resolve the lack of compliant robot-assisted hand motion and lack of intuitive user control in assistive and rehabilitation processes.

This proposed research aims to fill the above-mentioned gaps for current hand rehabilitation devices by developing a soft robotic glove that provides compliant assistance to bidirectional hand motion, coupled with intuitive user control.

In the short term, the robotic glove will likely enhance the patients' hand flexion-extension range of motion and improve the neuro-motor control of the hand.

In the long term, the robotic glove will act as an adjunct to therapists, thereby raising productivity in the presence of growing manpower constraints and optimizing therapy time for the patients; this can potentially enhance recovery time and quality of life, as a result of improved hand mobility for common daily tasks.

DETAILED DESCRIPTION:
The investigators aim to develop a new bidirectional composite soft actuator that is capable of assisting in both hand flexion and extension. This new class of actuator will comprise of a flexion actuator component with its external bending patterns and dedicated pneumatic channel, and an embedded extension actuator component with its dedicated air-flow inlet. When pressurized air is introduced through the extension inlet, the extension actuator will inflate and stiffen, thereby assisting in hand extension. Moreover, when pressurized air is introduced through the flexion inlet, the flexion actuator will inflate and bend, thereby assisting in hand flexion.

These bidirectional actuators will be embedded onto each finger segment of a fabric glove, and air inflow into each of the bidirectional actuators can be controlled via a pump-valve control system. The pump-valve control system comprises a microcontroller, onboard power source, transceiver, motor pump, and flexion and extension control valves. Once the microcontroller receives a command signal to adopt a specific hand posture, it will send the postural command to the motor pump and the necessary flexion/extension control valves, thereby actuating the corresponding bidirectional soft actuators to assist the user's hand into the desired hand posture.

Aims:

Aim 1: The bidirectional myoelectric soft robotic glove may provide intuitive user-controlled robot-assisted hand grasping postures to the human user for achieving functional tasks. With the help of the glove system, participants may be more capable of achieving active daily living tasks.

Aim 2: The bidirectional myoelectric soft robotic glove may provide intuitive user-controlled robot-assisted hand grasping postures to the human user for rehabilitation purposes.

Hypothesis:

The central hypothesis is that a bidirectional myoelectric soft robotic glove will provide intuitive user-controlled robot-assisted hand grasping postures to the human user for achieving functional tasks more than no robot assistance.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 30-90 years regardless of lesion size, race
2. Stroke type: ischemic or haemorrhagic
3. Fugl-Meyer Assessment (FMA) of upper extremity impairment of 10-56 out of a maximum score of 66 on the Fugl-Meyer assessment scale
4. Able to comprehend and follow commands
5. Unilateral upper limb impairment

Exclusion Criteria:

1. Recurrent stroke
2. Unstable medical conditions or anticipated life expectancy of <1 year
3. History of severe depression or active psychiatric disorder
4. Severe spasticity (Modified Ashworth scale >2)
5. Poor skin condition

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Functional Assessment | Change from Baseline FMA score at 6 weeks.
  Fugl-Meyer Assessment (FMA) Upper Extremity (UE) Score, A total of 66 scores.
Functional Assessment | Change from Baseline ARAT score at 6 weeks.
  Action Research Arm Test (ARAT), A total of 57 scores.
Brain Imaging | Change from Baseline Imaging at 6 weeks.
  Functional Magnetic Resonance Imaging

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Yap HK, Lim JH, Nasrallah F, Yeow CH. Design and Preliminary Feasibility Study of a Soft Robotic Glove for Hand Function Assistance in Stroke Survivors. Front Neurosci. 2017 Oct 9;11:547. doi: 10.3389/fnins.2017.00547. eCollection 2017. PMID 29062267
- [Background] Koh TH, Cheng N, Yap HK, Yeow CH. Design of a Soft Robotic Elbow Sleeve with Passive and Intent-Controlled Actuation. Front Neurosci. 2017 Oct 25;11:597. doi: 10.3389/fnins.2017.00597. eCollection 2017. PMID 29118693